CLINICAL TRIAL: NCT05586620
Title: Comparative Study on 3 Snip Punctoplasty With and Without Mitomycine C in the Management of Punctual Stenosis or Occlusion
Brief Title: 3 Snip Punctoplasty With and Without Mitomycine C.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Principal investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3 Snip Punctoplasty
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Punctal Stenosis
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-snip punctoplasty (Active Comparator)
  Interventions: Procedure: 3-snip punctoplasty
- 3-snip punctoplasty with mitomycin C (Active Comparator)
  Interventions: Procedure: 3-snip punctoplasty and Mitomycin C

INTERVENTIONS:
Procedure: 3-snip punctoplasty — punctoplasty, more commonly known as watery eye surgery, is an ophthalmic surgical procedure performed to correct punctal stenosis (a condition that causes tears to overflow from the eyes) by widening the punctal opening to allow the tears to drain with ease.
  Arms: 3-snip punctoplasty
Procedure: 3-snip punctoplasty and Mitomycin C — punctoplasty, more commonly known as watery eye surgery, is an ophthalmic surgical procedure performed to correct punctal stenosis (a condition that causes tears to overflow from the eyes) by widening the punctal opening to allow the tears to drain with ease.
  Mitomycin C is a chemotherapeutic agent that acts by inhibiting DNA synthesis
  Arms: 3-snip punctoplasty with mitomycin C

SUMMARY:
Punctal stenosis is a progressive constriction of the puncta with resultant epiphora. One of the most effective treatment options is 1- to 4-snip punctoplasty combined with or without Mitomycin-C.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrence of punctal stenosis at the end of 1 month following punctal dilatation.

Exclusion Criteria:

* patients with associated lacrimal passage obstruction

Ages: 16 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Punctal patency | Baseline
  Punctum will be assessed by inspection of the lid by slitlamb examination, whither obstructed or not
Punctal patency | 1 week postoperative
  Punctum will be assessed by inspection of the lid by slitlamb examination, whither obstructed or not
Punctal patency | 1 month postoperative
  Punctum will be assessed by inspection of the lid by slitlamb examination, whither obstructed or not
Punctal patency | 3 months postoperative
  Punctum will be assessed by inspection of the lid by slitlamb examination, whither obstructed or not
Presence of Epiphora | Baseline
  It will be assessed by inspection of the lid by slitlamb examination.
Presence of Epiphora | 1 week postoperative
  It will be assessed by inspection of the lid by slitlamb examination.
Presence of Epiphora | 1 month postoperative
  It will be assessed by inspection of the lid by slitlamb examination.
Presence of Epiphora | 3 month postoperative
  It will be assessed by inspection of the lid by slitlamb examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt